CLINICAL TRIAL: NCT05259098
Title: "Sufentanil Sublingual Tablet System vs Intravenous Patient-Controlled Analgesia With Morphine: Postoperative Pain Control and Its Impact in Quality of Recovery
Brief Title: Morphine vs Sufentanil PCA: Same Same or Different?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Central do Funchal (Other)
Responsible Party: Principal Investigator, Ana isabel freitas amorim, Ana Isabel Freitas Amorim, Hospital Central do Funchal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35/2019
Record Dates: First submitted 2022-02-07; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Analgesia; Post Operative Pain; Patient Satisfaction; Chronic Pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative; Patient Satisfaction; Chronic Pain | interventions — Sufentanil; Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sufentanil Sublingual Tablet System (Experimental): Group treated with Sufentanil Sublingual Tablet System
  Interventions: Drug: Sufentanil Sublingual Tablet System
- Intravenous Patient-Controlled Analgesia with Morphine (Experimental): Group treated with intravenous Patient-Controlled Analgesia with Morphine
  Interventions: Drug: Intravenous Patient-Controlled Analgesia with morfine

INTERVENTIONS:
Drug: Sufentanil Sublingual Tablet System — Sufentanil Sublingual Tablet System is a sublingual opioid patient controlled analgesia system. It was used for postoperative analgesia after surgery associated with moderate to severe pain.
  Other Names: zalviso
  Arms: Sufentanil Sublingual Tablet System
Drug: Intravenous Patient-Controlled Analgesia with morfine — Intravenous Patient-Controlled Analgesia with morfine. It was used for postoperative analgesia after surgery associated with moderate to severe pain.
  Arms: Intravenous Patient-Controlled Analgesia with Morphine

SUMMARY:
Patient-controlled intravenous analgesia (PCA) has already proven its quality. However, with new strategies starting to emerge and the current concept of opioid sparing, it is a goal to find the optimal PCA strategy capable of improve patient satisfaction and, at the same time, individualize opioid dose.

In a prospected randomized study, it was compared the use of Sufentanil Sublingual PCA System with intravenous PCA Morphine in terms of postoperative pain control satisfaction, total dose of opioid required, adverse effects, impact on the quality of postoperative recovery and the incidence of postoperative chronic pain.

DETAILED DESCRIPTION:
In a prospected randomized study, it was compared the use of Sufentanil Sublingual PCA System (15mcg per tablet, 20 minutes lockout) with intravenous PCA Morphine based on 1mg morphine on-demand 10 minutes lockout and a baseline perfusion of 1mg/hour.

45 patients capable of comply a PCA regime submitted to total knee arthroplasty, total hip arthroplasty and abdominal hysterectomy were enrolled in the study. During the first 48 hours, it was accessed daily pain scores, PCA use, need for rescue therapy, adverse effects, global satisfaction as well as postoperative quality recovery. Brief Pain Inventory was performed before surgery and 4 months later.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed;
* Age superior to 18 years;
* Physical status according to the American Society of Anesthesiology (ASA) 1-3;
* Scheduled gynecological surgery: abdominal hysterectomy
* Scheduled orthopedic surgery: total knee arthroplasty or total hip arthroplasty.

Exclusion Criteria:

* Patient refusal to participate in the study;
* Age <18 years or legal dependence;
* Neurological or psychiatric pathology or altered state of consciousness that does not allow for the Patient Controlled Analgesia strategy;
* Documented drinking habits and/or consumption of illicit drugs;
* Patients tolerant to opioid therapy (use of >15 mg oral morphine or its equivalent per day for the last 3 months);
* Documented obstructive Sleep Apnea Syndrome (OSAS);
* Patients on long-term oxygen therapy;
* Intraoperative use of intrathecal morphine;
* Use of anesthetic techniques in order to provide postoperative analgesia (eg, epidural catheter; peripheral nerve block; infiltration of the surgical wound with local anesthetic).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain control | Evaluation at 24 hours and 48 hours after surgery
  Comparison between patient controlled analgesia with IV morphine and sublingual sufentanil in Numeric Rating Scale

SECONDARY OUTCOMES:
Adverse effects associated with analgesia | Evaluation at 24 hours and 48 hours after surgery
  Evaluation of adverse effects of the PCA systems: sedation using the Richamond Agitation Sedation Scale (RASS); hypoxemia without oxygen supplementation: mild to moderate (SpO2 90-93%) or severe (SpO2<90%); hypotension; nausea or vomiting; dyspepsia; itching
Total daily dose of opioid | Evaluation at 24 hours and 48 hours after surgery
  Evaluation of total daily dose of each drug
Patients satisfaction with analgesia | Evaluation at 24 hours and 48 hours after surgery
  Evaluation of patient satisfaction using a qualitative scale: "Poor"; "Average"; "Good"; "Excellent"
Impact of the treatment on the quality of postoperative recovery | Evaluation at 24 hours after surgery
  Evaluation of recovery with application of validated quality of recovery score (QoR-15) questionnaire
Incidence of postoperative chronic pain | 4 months after surgey
  Assessment to persistent postoperative pain by completing the Brief Pain Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Ana IPG Pereira, Medical, Principal Investigator — Hospital Central do Funchal
Locations (1):
- Hospital Central do Funchal, Funchal, Madeira, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF